CLINICAL TRIAL: NCT00115674
Title: Smoking Research With Incarcerated Females
Brief Title: To Examine Smoking Behavior of Prisoners - 1
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Cropsey, Associate Professor, University of Alabama at Birmingham
Other Study IDs: NIDA-15774-1; 5R01CA141663-03 (NIH); K23-15774-1
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Smoking Behavior
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to understand the smoking behavior of female incarcerated smokers and to determine how smokers differ from non-smokers on measures of substance abuse, personality, criminal history, and mental illness

ELIGIBILITY:
Inclusion Criteria:

* all smokers, non-smokers, and ex-smokers

Exclusion Criteria:

* inability to understand English and inability to be able to provide informed consent due to mental impairment

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult women incarcerated in a state prison in Virginia are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2002-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cropsey, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Cropsey KL, Kristeller JL. Motivational factors related to quitting smoking among prisoners during a smoking ban. Addict Behav. 2003 Aug;28(6):1081-93. doi: 10.1016/s0306-4603(02)00230-7. PMID 12834652
- [Background] Cropsey K, Eldridge GD, Ladner T. Smoking among female prisoners: an ignored public health epidemic. Addict Behav. 2004 Feb;29(2):425-31. doi: 10.1016/j.addbeh.2003.08.014. PMID 14732432
- [Background] Haller DL, Miles DR, Cropsey KL. Smoking stage of change is associated with retention in a smoke-free residential drug treatment program for women. Addict Behav. 2004 Aug;29(6):1265-70. doi: 10.1016/j.addbeh.2004.03.029. PMID 15236833
- [Background] Cropsey KL, Kristeller JL. The effects of a prison smoking ban on smoking behavior and withdrawal symptoms. Addict Behav. 2005 Mar;30(3):589-94. doi: 10.1016/j.addbeh.2004.07.003. PMID 15718077